CLINICAL TRIAL: NCT03935360
Title: External Validation of a Prognostic Risk Score for Safe Discharge Among Patients With Lower Gastrointestinal Bleeding: A Prospective Multi-centre Cohort Study
Brief Title: Oakland-Jairath Score Validation
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Western University, Canada (Other); Université de Montréal (Other); University of Alberta (Other); McGill University (Other); University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: 113116
Record Dates: First submitted 2019-04-30; First posted 2019-05-02 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Lower Gastrointestinal Bleeding
Keywords: lower gastrointestinal bleeding; external validation; prognostic risk score; safe discharge; multi-centre cohort study; obscure gastrointestinal bleeding; hospital presentation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Oakland-Jairath Risk Score — Oakland and Jairath developed a clinical prediction rule for safe discharge among patients with LGIB using data from their UK National Audit. They defined safe discharge as the absence of rebleeding, blood transfusion, need for endoscopic/radiologic/surgical intervention for hemostasis, readmission with LGIB, and death and developed a seven variable risk score: age, sex, previous history of LGIB admission, presence of blood on digital rectal exam, heart rate, systolic blood pressure, and hemoglobin. Using a cut-off score ≤8, they reported excellent discrimination (AUC 0.84, 95% CI 0.82-0.86), good calibration, and a 95% probability of safe discharge.

SUMMARY:
Lower gastrointestinal bleeding (LGIB) is a common presentation in the Emergency Room. It can deteriorate into severe adverse event. However some are discharged before these events occur. The Oakland-Jairath score was developed to help determine which patients can be safely discharged and which should be admitted from the ER to the hospital. The score did well in its development, but now needs to be externally validated by other independent cohorts. The limitations of the first study will be addressed in our study. The goal of this study is to perform the first prospective, multi-centered, external validation of the Oakland-Jairath risk score on an independent and diverse population who present to the emergency room with LGIB.

DETAILED DESCRIPTION:
Of critical importance in the approach to care of these patients is differentiating the majority of people who can be safely discharged for outpatient management from those who are at risk for serious adverse events and require hospitalization. Recently, Oakland and Jairath developed a clinical prediction rule for safe discharge among patients with LGIB using data from their UK National Audit. The next step in the development of a clinical prediction rule is external validation in independent cohorts. Measures of predictive accuracy for risk scores, such as the AUC, are overly optimistic when calculated from the derivation cohort from which the risk score was derived. Therefore, it is essential to evaluate its performance using independent and diverse validation cohorts. Thus, the goal of this study is to perform the first prospective, multi-centered, external validation of the Oakland-Jairath risk score on an independent and diverse population who present to the emergency room with LGIB. This is a prospective multi-centre observational study to externally validate the Oakland-Jairath LGIB risk score, herein referred to simply as the "risk score".

Consecutive patients presenting to hospital over a 6 month period will have their risk score calculated and followed for the development of an adverse outcome over a 28 day period. The risk score will be determined for research purposes only but will be shared with the treating physician if requested as the details of the risk score itself is within the public domain. Patients will be eligible regardless of discharge status and all admission decisions will be made solely by the treating physicians. To increase the diversity of the validation cohort, increase generalizability, and hasten recruitment, the study will be conducted at 4 centres: Western University, University of Alberta, University of Montreal, and McGill University.

ELIGIBILITY:
Inclusion Criteria:

1. Presenting complaint of LGIB, defined as any of the following:

1. Bright red blood per rectum
2. Maroon coloured stool
3. Criteria A and B applies regardless if the blood is seen without stool, with stool of any consistency, or only on the toilet paper

Exclusion Criteria:

1. Age ≤ 18
2. Hematemesis, defined as bright blood or coffee ground emesis
3. Patients who developed LGIB while already admitted to hospital for any reason
4. Patients transferred between hospitals
5. Failure to obtain informed consent
6. Occult bleeding, defined as the presence of a positive FOBT/FIT or iron deficiency anemia in the absence of bright red blood per rectum or maroon coloured stool
7. Perceived inability to contact the subject by telephone or e-mail for the 28 day follow up assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any adult person who presents with lower gastointestinal bleeding as defined by: bright red blood per rectum, and/or maroon coloured stool.
Sampling Method: Probability Sample
Enrollment: 344 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2024-03-02 (Actual); Study Completion 2024-03-02 (Actual)

PRIMARY OUTCOMES:
Discrimination of the Oakland-Jairath score for predicting safe discharge | 28 days after enrollment
  Discrimination, defined as the ability of the prediction model to differentiate between those who develop and do not develop the outcome event of interest, as measured by the c-statistic, and calibration, defined as the agreement between predicted and observed outcomes, measured by a calibration plot, of the Oakland-Jairath score for predicting safe discharge, defined as the absence of ALL of the following:
  i. Rebleeding, defined as [additional blood transfusions] or [a further decrease in hematocrit concentration of 20% or more], both after 24h clinical stability ii. Readmission for LGIB within 28 days iii. Red blood cell transfusion iv. Therapeutic intervention for hemostasis (endoscopic/IR/surgery) v. Death within 28 days

SECONDARY OUTCOMES:
Discrimination of the Oakland-Jairath score compared to pre-existing LGIB risk scores | 28 days after enrollment
  Measured by the c-statistic and compared using the DeLong test The scale is Oakland & Jairath score for the prediction of safe discharge after LGIB. There are seven variables that are scored. Having a lower score in all variables and overall represents a better outcome for a safe discharge after LGIB.
  Age: <40 = 0; 40-69 =1; ≥70 =2 Sex: F = 0; M =1 Previous LGIB admission: No = 0; Yes = 1 DRE findings: No blood = 0; Blood = 1 Heart rate (bpm): ≤70 = 0; 70-89= 1; 90-109= 2; ≥110 = 3 Systolic blood pressure (mmHg): 50-89 = 5; 90-119 = 4; 120-129 = 3; 130-159 = 2; ≥160 = 0 Hemoglobin (g/dL): 36-69 = 22; 70-89 = 17; 90-109 = 13; 110-129 = 8; 130-159 = 4; ≥160 = 0
  Total with variables added together that translates to the probability of safe discharge:
  0-2 = 0.99; 3 = 0.98; 4 = 0.97; 5-7 = 0.96; 8 = 0.95; 9 = 0.93; 10 = 0.91; 11 = 0.89; 12-13 = 0.87-0.89; 14-15 = 0.77-0.81; 16-17 = 0.67-0.72; 18-20 = 0.50-0.62; 21-23 = 0.33-0.45; 24-26 = 0.20-0.28; 27-29 = 0.11-0.16; ≥30 = <0.1
Discrimination of the Oakland-Jairath score compared to traditional UGIB risk scores | 28 days after enrollment
  Measured by the c-statistic and compared using the DeLong test The scale is Oakland & Jairath score for the prediction of safe discharge after LGIB. There are seven variables that are scored. Having a lower score in all variables and overall represents a better outcome for a safe discharge after LGIB.
  Age: <40 = 0; 40-69 =1; ≥70 =2 Sex: F = 0; M =1 Previous LGIB admission: No = 0; Yes = 1 DRE findings: No blood = 0; Blood = 1 Heart rate (bpm): ≤70 = 0; 70-89= 1; 90-109= 2; ≥110 = 3 Systolic blood pressure (mmHg): 50-89 = 5; 90-119 = 4; 120-129 = 3; 130-159 = 2; ≥160 = 0 Hemoglobin (g/dL): 36-69 = 22; 70-89 = 17; 90-109 = 13; 110-129 = 8; 130-159 = 4; ≥160 = 0
  Total with variables added together that translates to the probability of safe discharge:
  0-2 = 0.99; 3 = 0.98; 4 = 0.97; 5-7 = 0.96; 8 = 0.95; 9 = 0.93; 10 = 0.91; 11 = 0.89; 12-13 = 0.87-0.89; 14-15 = 0.77-0.81; 16-17 = 0.67-0.72; 18-20 = 0.50-0.62; 21-23 = 0.33-0.45; 24-26 = 0.20-0.28; 27-29 = 0.11-0.16; ≥30 = <0.1

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sey, MD, Principal Investigator — Lawson Research; Western University
Locations (6):
- Canada (6):
  - University of Alberta Hospital, Edmonton, Alberta
  - Health Science Centre, Winnipeg, Manitoba
  - Nova Scotia Health - Victoria General Site, Halifax, Nova Scotia
  - London Health Sciences Centre, London, Ontario
  - Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No